CLINICAL TRIAL: NCT01879527
Title: A Randomized, Placebo-Controlled, Double-Blind, Phase IIa Study of Amiloride in the Treatment of Acute Autoimmune Optic Neuritis
Brief Title: Amiloride Hydrochlorothiazide as Treatment of Acute Inflammation of the Optic Nerve
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Fritz Leutmezer, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SSP-2; 2012-005113-39 (EudraCT Number)
Record Dates: First submitted 2013-06-13; First posted 2013-06-18 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Optic; Neuritis, With Demyelination
MeSH Terms: conditions — Neuritis | interventions — amiloride, hydrochlorothiazide drug combination; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amiloride hydrochlorothiazide (Active Comparator): 5,68 mg Amiloridhydrochloride 2H20 (analogue 4,32 mg Amilorid) und 50 mg Hydrochlorothiazid. Trade name of the agent: Amilostad HCT 5/50mg tablets Manufacturer: Stada initial dose: 1 x 5/50mg once daily target dose: 2 x 5/50mg once daily Patients will be provided with capsules (size 00) containing one tablet of study medication and instructed to take these capsules once daily in the morning together with breakfast. Visit 2 will be scheduled one week after baseline and at visit 2 patients will be provided with capsules containing two tablets of study medication
  Interventions: Drug: Amiloride hydrochlorothiazide
- Sugar pill (Placebo Comparator): Patients will be provided with capsules (size 00) containing sugar and instructed to take these capsules once daily in the morning together with breakfast.
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Amiloride hydrochlorothiazide — Blinding will be done by over-encapsulating amiloride HCT tablets and providing corresponding placebo capsules.Patients will be provided with capsules (size 00) containing one tablet of study medication (Amilostad HCT 5/50mg tablet or placebo) and instructed to take these capsules once daily in the morning together with breakfast. Visit 2 will be scheduled one week after baseline and at visit 2 patients will be provided with capsules containing two tablets of study medication. This maintenance dose will not be changed throughout the remaining study period. Placebo will be administered in the exact same manner.
  Other Names: Marketing Authorisation number: 1-22734; Trade name: Amilostad HCT
  Arms: Amiloride hydrochlorothiazide
Drug: Sugar pill — containing placebo
  Other Names: placebo
  Arms: Sugar pill

SUMMARY:
Following acute inflammation of the optic nerve region, as commonly seen in multiple sclerosis patients, the optic nerve often undergoes atrophy, thus representing permanent damage. Data from animal studies suggest that amiloride may prevent this process. The aim of this study is to assess a potential neuroprotective effect of amiloride in acute autoimmune inflammation of the optic nerve region.

DETAILED DESCRIPTION:
Recent studies have shown that the acid-sensing ion channel 1 (ASIC1) contributes to the axonal degeneration in CNS lesions Physiologically, ASIC1 has been described as a postsynaptic proton receptor on hippocampal neurons influencing the intracellular Ca2+ concentration. In MS, ASIC1 seems to activate under acidic conditions predominating in the inflammatory CNS lesions leading to a Na+ and Ca2+ overload and consecutive damage and apoptosis of axons. Consecutively, in a MS mousemodel axonal damage was significantly less pronounced after administering amiloride, a clinically safe blocker of ASICs. So ASIC1 seems to play a major role in axonal degeneration in MS. To our knowledge no clinical studies have tested those promising in vitro results in humans so far.

Only one retrospective registry-based cohort study was performed. This study showed no difference in the risk of incident MS or hospitalization and death among MS patients using amilorid compared to those using thiazide diuretics. However, this study has numerous limitations with respect to it's retrospective designone and the fact that amilorid users were at the vast majority older individuals. Such a late stage of the MS course does not seem to be the best window of opportunity for interventions with neuroprotective agents. Moreover, death may be a too multifactorial parameter to correspond with axonal damage alone. Consequently, a more sensitive parameter for axonal damage in MS is needed to test the impact of amiloride on neuroprotection and repair.Based on the findings described above we intend to assess the potential neuroprotective effect of amiloride hydrochlorothiazide (Amilostad HCT®) in patients with optic neuritis (ON), which has already been demonstrated in a mouse model. ON is one of the most common manifestations of MS and has already been proven appropiate to test neuroprotective agents.

ELIGIBILITY:
Inclusion Criteria:

Patients between 18 and 50 years of age with a first episode of optic neuritis (ON) and a visual acuity decreased to <0,6 will be eligible for inclusion in the study. Diagnosis of ON has to be confirmed by an ophthalmologist. Onset of symptoms has to be within 10 days prior to inclusion into the study

Exclusion Criteria:

* Known allergy or hypersensitivity to amilostad HCT or any of its ingredients
* Known allergy or hypersensitivity to other sulphonamide-derived drugs
* Impaired renal function or any known renal disease
* Intake of other potassium-conserving diuretics
* Intake of potassium supplements or a special potassium rich diet
* Intake of spironolactone or triamterene
* Moderate to severe hepatic failure
* Morbus Addison
* Known hypercalcaemia
* Intake of lithium therapy
* Blood urea > 10mmol/l
* Diabetes mellitus
* History of ON or any other ocular disease (affected as well as unaffected eye)
* Pregnancy or lactation period
* Treatment with corticosteroids or amiloride within 30 days prior to the inclusion into the study
* Use of any immunomodulatory or immunosuppressive agents anytime in the past
* Dearrangement of serum sodium or potassium levels on the lab

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Change in thickness of retinal nerve fiber layer (RNFL) | Baseline versus follow-up at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fritz Leutmezer, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Neurology, Vienna, Vienna, Austria